CLINICAL TRIAL: NCT00071721
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of Valproate to Attenuate the Progression of Alzheimer's Disease (AD)
Brief Title: Valproate in Dementia (VALID)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alzheimer's Disease Cooperative Study (ADCS) (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IA0043; 1RC2AG036535 (NIH); IND 67,222; ADCS Protocol ADC-022-VN
Record Dates: First submitted 2003-10-29; First posted 2003-10-31 (Estimated); Results first posted 2010-10-20 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer disease; Agitation; Psychosis
MeSH Terms: conditions — Alzheimer Disease; Psychomotor Agitation; Psychotic Disorders | interventions — Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Valproate
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Valproate — 250mg tablets beginning with one daily for one week, then two daily for one week, then titrated according to body weight and tolerability to achieve 10-12 mg/kg daily for 2 years, followed by a 2-month washout
  Other Names: Depakene, Depakote
  Arms: 1
Drug: Placebo — Placebo tablets beginning with one daily and increasing according to weight and perceived tolerability concerns for two years, followed by a 2-month washout
  Arms: 2

SUMMARY:
The purpose of this trial is to demonstrate whether valproate therapy delays the emergence of agitation and/or psychosis in outpatients with probable Alzheimer's disease (AD) who have not experienced agitation and psychosis in their illness. A secondary aim is to determine whether valproate therapy delays the progression of cognitive and functional measures of the illness. This trial will also assess the tolerability and safety of low-dose, long-term valproate therapy. Valproate, an anticonvulsant drug, was selected because of its possible symptomatic efficacy for agitation in AD, known safety profile in numerous clinical populations, and in view of recent data supporting its neuroprotective potential in AD.

DETAILED DESCRIPTION:
This study represents a novel clinical trial strategy designed to assess both prospective "prophylactic" therapy for psychopathology in Alzheimer's disease (AD) and to assess an approach that may alter several aspects of the pathophysiology of AD, and perhaps result in alteration of clinical progression of illness. Interpretation of these results will be supported by study of relevant biomarkers and imaging data. Valproate was selected because of its possible symptomatic efficacy for agitation in AD, known safety profile in numerous clinical populations, and in view of recent data supporting its neuroprotective potential in AD. The primary hypothesis is that chronic valproate administration to participants with AD who lack agitation and psychosis at baseline will delay the emergence of agitation and/or psychosis. An effect of this nature may have significant public health implications, for instance, by delaying institutionalization.

This is a randomized, placebo-controlled, double blind, multicenter 26-month trial of valproate therapy at a target dose of 10-12 mg/kg/day in 300 outpatients with mild to moderate Alzheimer's Disease (AD) who lack agitation and psychosis at baseline and since onset of illness. Participants will have regular clinic visits as well as telephone contacts for assessment of behavior, cognition, function, safety and tolerability. The chief secondary aim is to determine whether valproate administration to participants with AD will attenuate clinical progression of illness measured by a reduced rate of cognitive or functional decline. In addition, issues related to safety and tolerability with low-dose (10-12 mg/kg/day) therapy will be addressed. Biological specimens will be obtained to study markers selected for their relevance to the disease as well as the postulated mechanism of action of the valproate therapy. Magnetic resonance imaging (MRI) scans will be performed prior to experimental treatment and after one year in a subset of participants in order to address possible drug-placebo differences in brain volume measures.

Approximately 300 participants from 25-35 clinical trial centers in the United States will be enrolled. Participation will include men and women with a diagnosis of probable Alzheimer's disease, age 55 or older, weighing at least 40 kg (88.2 lbs.), residing in the community at baseline, Mini Mental State Examination (MMSE) 10-20 inclusive, who have not experienced agitation or psychosis since the onset of their illness and who do not require treatment with psychotropic medications with the exception of antidepressants used only for treatment of depressive symptoms and limited use of sedatives for sleep. Participants, their relatives, guardians or authorized representatives and informants will be given ample opportunity to inquire about details of the study. Informed consent forms covering consent for the trial itself as well as the genetic research and biological sample storage and MRI scans will be provided to protect the patient's rights and confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Probable AD by National Institute of Neurological Disorders and Stroke (NINDS)-Alzheimer's Disease and Related Disorder Association (ADRDA) criteria.
* Males or females.
* > 55 and < 90 years of age.
* Weight > 40 kg (88.2 lbs.).
* Residing in the community at Screen and Baseline. Participants may reside in assisted living facilities, but not in long-term care nursing facilities or assisted living facilities that provide intensive support for people with dementia nor may they reside in a secure unit necessary for behavioral management.
* Mini Mental State Examination (MMSE) at Screen and Baseline 12-20 inclusive.
* Computed tomography (CT) or magnetic resonance imaging (MRI) since onset of dementia consistent with the diagnosis of probable AD. Single lacunes in non-critical areas and non-specific white matter changes that are interpreted as age-related are not grounds for exclusion. Any ambiguous scan results must be reviewed with the Project Director.
* Fluent in English or Spanish.
* Supervision available for study medication.
* Study partner to accompany subject to all visits.
* Study partner must have in-person contact with the participant > 2 days/week.
* Able to ingest oral medication.
* Total Neuropsychiatric Inventory (NPI) score for previous 4 weeks < 8 at Screening, and for the period between Screening and Baseline.
* NPI item score for the items assessing delusions, hallucinations, agitation/aggression all greater than or equal to 1 for 4 weeks prior to Screening (less than once/week and mild severity at most) and for the period between Screening and Baseline.
* Scores of greater than or equal to 1 for items rating delusions, hallucinations, and agitation/aggression taken from the NPI, modified to assess these features since onset of illness. This will be derived from a second interview with the modified NPI. (Agitation/psychosis during episodes of delirium are not considered exclusionary.).

Exclusion Criteria:

Exceptions to these criteria may be considered on a case-by-case basis at the discretion of the Project Director:

* Non-AD dementia.
* Females of child-bearing potential.
* Residence in a long-term care facility or equivalent at Baseline.
* Presence or previous history of agitation or psychosis requiring active psychotropic medication since the illness began.
* History of clinically significant stroke.
* Current evidence or history in past two years of: focal brain lesion, head injury with loss of consciousness or Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) criteria for any major psychiatric disorder including psychosis, major depression, bipolar disorder, alcohol or substance abuse.
* Sensory impairment that would prevent subject from participating in or cooperating with the protocol.
* Medical contraindications to study participation.
* Use of another investigational agent within two months prior to Screening.
* Evidence of any significant clinical disorder or laboratory finding that renders the subject unsuitable for receiving an investigational new drug including clinically significant or unstable hematologic, hepatic, cardiovascular, pulmonary, gastrointestinal, endocrine, metabolic, renal, or other systemic disease or laboratory abnormality.
* Clinical contraindication to the use of valproate (e.g., known hypersensitivity or allergic reactions, severe neutropenia, severe hepatic disease, or urea cycle disorder. A urea cycle disorder should be considered in patients with history of unexplained encephalopathy following protein meals, or family history of urea cycle disorder).
* History of seizure within past 5 years prior to Screening.
* Platelet count < 100,000/mm^3.
* International Normalized Ratio (INR) > 1.2 or partial thromboplastin time (PTT) > 40 seconds.
* Active neoplastic disease. Exceptions: skin tumors other than melanoma are not excluded; patients with stable prostate cancer may be included at the discretion of the Project Director; women who have been treated for breast cancer and have no metastases and whose survival is expected to exceed 2 years may be considered for inclusion on a case-by-case basis in consultation with the Project Director; patients with purely localized bladder wall cancers may be included at the discretion of the Project Director.

Excluded Medications:

* Use of psychotropics for treatment of agitation or psychosis. Antidepressants used in stable doses for 3 months prior to Screening to treat depression or anxiety, but not agitation, will be permitted. Low dose sedatives for sleep, but not agitation, will be permitted. Cholinesterase inhibitors used in stable doses for at least 3 months prior to Screening are permitted.
* Regular use of narcotic analgesics within 3 months of Screening.
* Anti-parkinsonian medications (e.g. levodopa, selegiline, pergolide, bromocriptine, pramipexole) within 2 months of Screening.
* Use of drugs with significant central anticholinergic or antihistaminic effects (eg, benztropine, trihexyphenidyl, dicyclomine, diphenhydramine, cyproheptadine, diphenoxylate, hydroxyzine, meclizine, prochlorperazine, promethazine) within 2 months of Screening.
* Use of other investigational drug studies within two months prior to Screening.
* Use of other anticonvulsants within 5 years prior to Screening.
* Use of zidovudine at any time.
* Use of tricyclic antidepressants within 1 month prior to Screening.
* Regular use of high doses of salicylates at Screening (> 1,300 mg/d).
* Vitamin E > 2,100 IU/d within 1 month prior to Screening.
* Warfarin use is permitted when approved by the Project Director and INR and PTT criteria are met.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2003-10; Primary Completion 2009-02 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Tariot, MD, Study Director — University of Rochester Medical Center, Departments of Psychiatry, Medicine, and Neurology, and the Center for Aging and Developmental Biology
Locations (46):
- United States (46):
  - Sun Health Research Institute, Sun City, Arizona
  - University of Arizona, Tucson, Arizona
  - University of California, Irvine, Irvine, California
  - University of California, ADRC, San Diego, La Jolla, California
  - VA Healthcare System Long Beach, Long Beach, California
  - University of Southern California, Los Angeles, California
  - University of California ADRC, Los Angeles, California
  - University of California, LA (Olive View), Los Angeles, California
  - Pacific Research Network, San Diego, California
  - Stanford University, VA Aging Clinical Research Center, Stanford, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Howard University, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Florida
  - Wein Center, Mount Sinai Medical Center, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Byrd Institute, Tampa, Florida
  - Premier Research Institute, West Palm Beach, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Southern Illinois University, Springfield, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Kansas, Kansas City, Kansas
  - Lahey Clinic, Research Neurology, Burlington, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Saint Mary's Health Care, Grand Rapids, Michigan
  - St. Louis University, St Louis, Missouri
  - University of Nevada, Las Vegas, Nevada
  - Albany Medical Center, Albany, New York
  - Dent Neurologic Institute, Amherst, New York
  - New York University Medical Center, New York, New York
  - Columbia University, New York, New York
  - Global Research and Consulting, Olean, New York
  - University of Rochester, Rochester, New York
  - Syracuse VA Medical Center, Syracuse, New York
  - North East Ohio Health Services, Beachwood, Ohio
  - Case Western Reserve University, University Hospitals of Cleveland, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Brown University, Memorial Hospital of Rhode Island, Providence, Rhode Island
  - Medical University of South Carolina-Columbia, Columbia, South Carolina
  - Medical University of South Carolina-Florence, Florence, South Carolina
  - Medical University of South Carolina, North Charleston, South Carolina
  - Psychiatric Consultants, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Southwestern Vermont Medical Center, Bennington, Vermont
  - University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Background] Tariot PN, Loy R, Ryan JM, Porsteinsson A, Ismail S. Mood stabilizers in Alzheimer's disease: symptomatic and neuroprotective rationales. Adv Drug Deliv Rev. 2002 Dec 7;54(12):1567-77. doi: 10.1016/s0169-409x(02)00153-9. PMID 12453674
- [Background] Manji HK, Moore GJ, Rajkowska G, Chen G. Neuroplasticity and cellular resilience in mood disorders. Mol Psychiatry. 2000 Nov;5(6):578-93. doi: 10.1038/sj.mp.4000811. PMID 11126389
- [Background] Chen G, Huang LD, Jiang YM, Manji HK. The mood-stabilizing agent valproate inhibits the activity of glycogen synthase kinase-3. J Neurochem. 1999 Mar;72(3):1327-30. doi: 10.1046/j.1471-4159.2000.0721327.x. PMID 10037507
- [Derived] Tariot PN, Schneider LS, Cummings J, Thomas RG, Raman R, Jakimovich LJ, Loy R, Bartocci B, Fleisher A, Ismail MS, Porsteinsson A, Weiner M, Jack CR Jr, Thal L, Aisen PS; Alzheimer's Disease Cooperative Study Group. Chronic divalproex sodium to attenuate agitation and clinical progression of Alzheimer disease. Arch Gen Psychiatry. 2011 Aug;68(8):853-61. doi: 10.1001/archgenpsychiatry.2011.72. PMID 21810649

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Valproate | Placebo
Started | 153 | 160
Completed | 81 | 69
Not Completed | 72 | 91

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Valproate | Placebo | Total
Number analyzed (Participants) | 153 | 160 | 313
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.9 (8.2) | 76.6 (7.4) | 75.7 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 101 | 184
  Male | 70 | 59 | 129
Region of Enrollment [Number; unit: participants]
  United States | 153 | 160 | 313
ADAScog [Mean (Standard Deviation); unit: Units on a scale] — Alzheimer's Disease Assessment Scale, cognitive sub-scale in points per year (ADAS-cog) is a psychometric measure sensitive to change in mild to moderate AD. The range of this instrument is 0 to 70 with higher numbers indicating greater impairment.
  Units on a scale | 29.4 (8.9) | 30.1 (9.8) | 29.8 (9.4)
ADCS-ADL [Mean (Standard Deviation); unit: Units on a scale] — Alzheimer's Disease Cooperative Study Activities of Daily Living Score (ADCS-ADL) is a structured questionnaire about activities of daily living, administered to the subject's caregiver/study partner. The range of this instrument is 0 to 78 with lower numbers indicating greater impairment.
  Units on a scale | 56.9 (11.8) | 54.9 (13) | 55.9 (12.4)
CDR-SOB [Mean (Standard Deviation); unit: Units on a scale] — Clinical Dementia Rating, Sum of Boxes (CDR-SOB) is a global rating of dementia severity based on the clinician's interpretation of the history and examination. The range of this instrument is 0 to 18 with higher numbers indicating greater impairment.
  Units on a scale | 7.1 (2.7) | 7.5 (3.1) | 7.3 (2.9)
CMAI [Mean (Standard Deviation); unit: Units on a scale] — The Cohen-Mansfield Agitation Inventory (CMAI) is a 29-item caregiver rating questionnaire for the assessment of agitation in older persons. It includes descriptions of 29 agitated behaviors, each rated on a 7-point scale of frequency. The range of this instrument is 29 to 203 with higher numbers indicating greater impairment.
  Units on a scale | 10.9 (8.9) | 11.9 (10.4) | 11.4 (9.7)
NPI [Mean (Standard Deviation); unit: Units on a scale] — The Neuropsychiatric Inventory (NPI) quantifies behavioral changes in dementia, including depression, anxiety, psychosis, agitation, sleep change, appetite change, and others. This is a structured questionnaire administered to the subject's caregiver/study partner. The range of this instrument is 0 to 120 with higher numbers indicating greater impairment.
  Units on a scale | 2.6 (2.6) | 3.1 (2.6) | 2.9 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Presence of Agitation and/or Psychosis Measured by the Neuropsychiatric Inventory (NPI) Combined With an Assessment of the Clinical Significance of Behavioral Change Rated by the Study Clinician
Description: NPI quantifies behavioral changes in dementia, including depression, anxiety, psychosis, agitation, and others. This is a questionnaire administered to the subject's study partner. The range of this instrument is 0 to 120 with higher numbers indicating greater impairment. To determine whether or not psychosis or agitation is present, there is no cutoff score but is based on the clinician's judgment. In the NPI, the subject responds to 'Yes' or 'No' questions. Then it is determined how often psychosis or agitation occurs and if it is mild, moderate or severe.
Time Frame: 24 months
Measure: Number; unit: Participants
Arm/Group | Valproate | Placebo
Number analyzed (Participants) | 153 | 160
Participants | 25 | 29
Statistical Analysis 1: Comparison: Valproate vs Placebo; Test type: Superiority or Other; p = 0.88, Cox Proportional Hazards; Cox Proportional Hazard = 0.958

2. Secondary Outcome: Cognitive Performance Assessed by the Alzheimer's Disease Assessment Scale-cognitive Subtest (ADAS-cog)
Description: Alzheimer's Disease Assessment Scale, cognitive sub-scale in points per year (ADAS-cog) is a psychometric measure sensitive to change in mild to moderate AD. The range of this instrument is 0 to 70 with higher numbers indicating greater impairment.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Valproate | Placebo
Number analyzed (Participants) | 153 | 160
Units on a scale | 42.3 (14.3) | 41.9 (14.4)

3. Secondary Outcome: Functional Performance Assessed by the Alzheimer's Disease Cooperative Study Activities of Daily Living (ADCS-ADL) Inventory
Description: Alzheimer's Disease Cooperative Study Activities of Daily Living Score (ADCS-ADL) is a structured questionnaire about activities of daily living, administered to the subject's caregiver/study partner. The range of this instrument is 0 to 78 with lower numbers indicating greater impairment.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Valproate | Placebo
Number analyzed (Participants) | 153 | 160
Units on a scale | 35.1 (20.3) | 41.0 (14.81)

4. Secondary Outcome: Global Severity of Dementia Using the CDR Sum of Boxes
Description: Clinical Dementia Rating, Sum of Boxes (CDR-SOB) is a global rating of dementia severity based on the clinician's interpretation of the history and examination. The range of this instrument is 0 to 18 with higher numbers indicating greater impairment.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Valproate | Placebo
Number analyzed (Participants) | 153 | 160
Units on a scale | 12.0 (4.1) | 11.5 (3.7)

5. Secondary Outcome: Agitation Measured by the Cohen-Mansfield Agitation Inventory (CMAI), Community Version
Description: The Cohen-Mansfield Agitation Inventory (CMAI) is a 29-item caregiver rating questionnaire for the assessment of agitation in older persons. It includes descriptions of 29 agitated behaviors, each rated on a 7-point scale of frequency. The range of this instrument is 29 to 203 with higher numbers indicating greater impairment.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Valproate | Placebo
Number analyzed (Participants) | 153 | 160
Units on a scale | 10.6 (11.6) | 12.1 (10.9)

6. Secondary Outcome: Participant's Clinical Condition or Endpoint Assessed With the ADCS-Clinical Global Impression of Change (ADCS-CGIC)
Description: ADCS-Clinical Global Impression of Change (ADCS-CGIC) provides a means to reliably assess global change from baseline. It provides a semi-structured format to allow clinicians to gather necessary clinical information from both the participant and informant, in order to make an overall impression of clinical change. The range of this instrument is 1 to 7 with lower numbers indicating improvement and higher numbers indicating a worsened state.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Valproate | Placebo
Number analyzed (Participants) | 153 | 160
Units on a scale | 5.7 (0.9) | 5.5 (1.1)

ADVERSE EVENTS:
Arm/Group | Valproate | Placebo
Serious Adverse Events (participants affected / at risk) | 51/153 | 62/160
Other Adverse Events (participants affected / at risk) | 145/153 | 151/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valproate (N=153) | Placebo (N=160)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (4) | 1 (2)
Bladder repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast reconstruction (Surgical and medical procedures) | 0 (0) | 1 (1)
Breast swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (2)
Cardiac pacemaker replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Cerebral artery occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 3 (3) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 4 (4)
Coordination abnormal (Nervous system disorders) | 0 (0) | 1 (1)
Death (General disorders) | 5 (5) | 7 (7)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Drug toxicity (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 6 (6) | 9 (10)
Femoral hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gallbladder operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hepatic mass (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Hospitalisation (Surgical and medical procedures) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Joint arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 2 (2) | 0 (0)
Knee operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Leg amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Lesion excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Lethargy (Psychiatric disorders) | 0 (0) | 1 (1)
Listeriosis (Infections and infestations) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mental disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Oesophageal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 6 (6)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Postoperative infection (Infections and infestations) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Vascular disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Subdural haematoma (Nervous system disorders) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Subdural haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 4 (4) | 2 (2)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (5) | 3 (3)
Uterine prolapse repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Ventriculo-peritoneal shunt (Surgical and medical procedures) | 0 (0) | 1 (1)
Whole blood transfusion (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valproate (N=153) | Placebo (N=160)
Abdominal discomfort (Gastrointestinal disorders) | 16 (19) | 13 (13)
Agitation (Psychiatric disorders) | 43 (50) | 54 (74)
Anxiety (Psychiatric disorders) | 24 (29) | 38 (47)
Apathy (Psychiatric disorders) | 9 (9) | 9 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 (21) | 12 (14)
Asthenia (General disorders) | 48 (52) | 35 (37)
Back pain (Musculoskeletal and connective tissue disorders) | 21 (21) | 20 (20)
Bronchitis (Infections and infestations) | 7 (8) | 5 (6)
Chest pain (General disorders) | 7 (9) | 8 (8)
Confusional state (Psychiatric disorders) | 76 (114) | 79 (111)
Constipation (Gastrointestinal disorders) | 26 (28) | 13 (16)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (24) | 18 (22)
Crying (Psychiatric disorders) | 23 (27) | 22 (24)
Decreased appetite (Metabolism and nutrition disorders) | 8 (9) | 7 (8)
Delusion (Psychiatric disorders) | 10 (11) | 14 (20)
Depressed mood (Psychiatric disorders) | 35 (37) | 23 (26)
Depression (Psychiatric disorders) | 18 (19) | 10 (11)
Diarrhoea (Gastrointestinal disorders) | 38 (45) | 19 (24)
Disturbance in attention (Nervous system disorders) | 40 (40) | 39 (39)
Dizziness (Nervous system disorders) | 23 (25) | 30 (36)
Dry mouth (Gastrointestinal disorders) | 16 (16) | 15 (15)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 (20) | 9 (9)
Faecal incontinence (Gastrointestinal disorders) | 8 (8) | 5 (5)
Fall (Injury, poisoning and procedural complications) | 54 (85) | 42 (86)
Gait disturbance (Nervous system disorders) | 51 (64) | 30 (35)
Hallucination (Psychiatric disorders) | 9 (11) | 5 (5)
Headache (Nervous system disorders) | 16 (19) | 13 (16)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4) | 9 (9)
Insomnia (Psychiatric disorders) | 20 (23) | 16 (18)
Joint swelling (Musculoskeletal and connective tissue disorders) | 14 (15) | 10 (12)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 28 (32) | 14 (14)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (12) | 11 (12)
Nasopharyngitis (Infections and infestations) | 11 (12) | 9 (13)
Nausea (Gastrointestinal disorders) | 14 (16) | 10 (11)
Oedema peripheral (General disorders) | 10 (12) | 7 (7)
Pollakiuria (Renal and urinary disorders) | 23 (25) | 17 (19)
Rash (Skin and subcutaneous tissue disorders) | 7 (7) | 15 (17)
Restlessness (Psychiatric disorders) | 28 (34) | 31 (39)
Somnolence (Psychiatric disorders) | 66 (80) | 46 (51)
Tremor (Nervous system disorders) | 44 (51) | 22 (23)
Urinary incontinence (Renal and urinary disorders) | 15 (18) | 15 (16)
Urinary tract infection (Infections and infestations) | 15 (19) | 17 (28)
Vision blurred (Eye disorders) | 10 (11) | 8 (8)
Vomiting (Gastrointestinal disorders) | 9 (10) | 7 (7)
Weight decreased (Investigations) | 11 (12) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No